CLINICAL TRIAL: NCT00419367
Title: Compassionate Use of Vorinostat (MK0683) for the Treatment of Patients With Advanced Cutaneous T-Cell Lymphoma
Brief Title: Compassionate Use of Vorinostat for the Treatment of Patients With Advanced Cutaneous T-Cell Lymphoma (0683-042)
Status: No longer available | Type: Expanded Access
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0683-042; MK0683-042; 2006_540; 2006-003879-12 (EudraCT Number)
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Lymphoma, T-Cell, Cutaneous
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

INTERVENTIONS:
Drug: Comparator: vorinostat — Each patient will receive open-label vorinostat 400 mg q.d. capsules. Treatment will continue until disease progression, intolerable toxicity, withdrawal of consent, or physician determines it is in best interest of patient to withdrawal.

SUMMARY:
In an effort to allow patients continued access to vorinostat outside of the base study, patients that are actively receiving study medication will discontinue from this study and receive vorinostat via another method supported by the SPONSOR (e.g. Named Patient Program (NPP)). For those institutions that do not allow receipt of an investigational therapy outside of a clinical trial, patients that are actively receiving study medication and

continue to meet eligibility will transition to an extension phase of the study and the base study will be closed.

The extension phase will begin as soon as the protocol amendment is implemented.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cutaneous T-cell lymphoma on or following two systemic therapies
* Female participants must have a negative serum pregnancy test within 3 days of the first dose of vorinostat
* Female participants must have finished menopause, or are surgically sterilized, or agree to use 2 adequate barrier methods of contraception
* Male participants must agree to use 2 adequate barrier methods of contraception
* To be treated on extension phase of study participant must have been treated on the base study for Protocol 042

Exclusion Criteria:

* Currently receiving any potential histone deacetylase (HDAC) inhibitor (e.g. valproic acid)
* Currently receiving any other systemic therapy for CTCL. Corticosteroids that are similar in strength to 20 mg of prednisone daily are permitted
* Pregnant or lactating
* Known allergy to any component of the study drug
* Eligible for any other study of vorinostat in CTCL patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC